CLINICAL TRIAL: NCT02410941
Title: Improving the Stewardship of Diagnostic Imaging Resources in Alberta Emergency Departments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Dr. Eddy S. Lang, Doctor, associate professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10007399
Record Dates: First submitted 2015-03-17; First posted 2015-04-08 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Brain Injuries; Pulmonary Embolism
Keywords: Randomized controlled trial; Practice management; tomography, x-ray computed/adverse effects; Clinical decision support; Computerized clinical decision support; Decision support systems, clinical; Health Expenditures; Physician's practice patterns; Unnecessary Procedures/economics; Physician's Practice Patterns/economics; Diffusion of innovation; Decision Support Models; Clinical Prediction Rules
MeSH Terms: conditions — Brain Injuries; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision-support for MTBI (Experimental): Clinical decision support will be provided on ordering CT scans for patients suspected to have Minor Traumatic Brain Injury (MTBI) to treating physicians randomized into this group. This arm will also serve as a control for the PE group.
  Interventions: Behavioral: Clinical decision support
- Decision-support for PE (Experimental): Clinical decision support will be provided on ordering CT scans for patients suspected to have Pulmonary Embolism (PE) to treating physicians randomized into this group. This arm will also serve as a control for the MTBI group.
  Interventions: Behavioral: Clinical decision support

INTERVENTIONS:
Behavioral: Clinical decision support — Establish evidence-based standardized clinical pathways implemented by local communities of practice focused on imaging utilization in ED settings as models of participatory research and integrated knowledge translation.

SUMMARY:
Utilization of diagnostic imaging in the Emergency Department has increased dramatically over the past two decades, driven by an increased availability of advanced imaging, legal pressures to exclude serious diagnoses in low-risk patients, patient expectations, and the tendency to associate more testing with a higher quality of care. However, this rise in the use of diagnostic imaging, particularly in low-risk patients, may not be taking into account the risk of radiation exposure to patients, or the impact on finite health system resources. The objective of this project is to improve the appropriateness of CT imaging in Alberta Emergency Departments by advancing awareness of, and adherence to, evidence-based guidelines for CT imaging of patients with mild traumatic brain injury (MTBI) and suspected pulmonary embolism (PE). These two clinical scenarios have been selected because of evidence of significant variation in imaging practices across Alberta, and the robust evidence base that exists to guide CT imaging decisions such as the Canadian CT Head Rule and the Pulmonary Embolism Rule Out Criteria.

DETAILED DESCRIPTION:
Background:

Imaging technology for the rapid diagnosis of medical conditions is an indispensable tool in the emergency department (ED). However, increasing and inappropriate use of costly and potentially dangerous imaging is a growing healthcare concern. The long-term health risks of radiation exposure, and the resources consumed by increased use, pose serious threats to the integrity of the investigators' health care system and the population at large. Computed tomography (CT) is frequently used in the emergency department setting to evaluate patients with mild traumatic brain injury (MTBI) and suspected pulmonary embolism (PE) to eliminate diagnostic uncertainty by either confirming or ruling out serious injury and illness. However, these tests are often used in lieu of alternate and safer strategies with equivalent accuracy and effectiveness. Fortunately, well-validated decision-support tools exist that can safely identify low risk patients who are unlikely to benefit from CT imaging, avoiding unnecessary diagnostic imaging and radiation exposure, and making better use of limited health system resources. However, decision-support is under-used in clinical practice, and research to optimize their uptake has yielded mixed results.

Study Objectives:

The investigators will conduct a cluster-randomized trial to evaluate whether the implementation of decision-support into standard clinical practice for ordering CTs will (a) decrease the number of CTs ordered, (b) increase the appropriateness of the CTs that are ordered (e.g. by increasing diagnostic yield but avoiding any missed diagnosis).

Scope:

The scope is to focus on two conditions for which validated decision-support exists: MTBI and PE.

These conditions were selected because internal AHS data shows significant variability (15-90%) in the ordering of CTs for patients presenting with these conditions, and because validated decision-support exists for these conditions (e.g. Canadian CT Head Rule, Well's Score, Pulmonary Embolism Rule-Out Criteria).

The scope includes all hospitals in Alberta with an ED and in-house CT. There are 17 of these hospitals in Alberta from Fort McMurray to Medicine Hat. The investigators have obtained operational approvals to conduct the researchers' study in all 17 hospitals from the Emergency Chief at each site, and from ED and Diagnostic Imaging leadership at the level of each Zone as well as the Province. The scope is limited to patients presenting to the ED.

Methods:

The study design is a cluster randomized trial. In the Calgary Zone, the investigators will randomize half of the investigators' ED physicians to receive decision-support for MTBI, and half to receive decision-support for PE.

Outside of the Calgary Zone, the investigators will randomize by site, so half of sites will receive decision-support for MTBI, and half will receive decision-support for PE. Each half of the randomization will serve as a control for the other group. The reason the investigators are randomizing by physician in the Calgary Zone is because the Computerized Physician Order Entry system in Calgary allows us to implement such a randomization, whereas outside of the Calgary Zone the heterogeneity of order entry systems does not make it feasible to randomize by physician, but it is feasible to randomize by site.

The implementation of decision-support for CT ordering will be mandatory and is supported by operational and clinical leadership. By integrating decision-support into the existing systems to order CTs, a physician (or site) randomized to MTBI or PE decision-support will have to consider those tools prior to ordering a CT. However, decision-support does not make decisions about who receives a CT; it merely provides additional information about how likely a CT is to be diagnostically useful. All decisions regarding diagnostic or therapeutic interventions are the sole responsibility of the physician in consultation with the patient. The primary outcomes measured by this study will be (a) the percentage of MTBI and PE patients receiving a CT scan, and (b) the "appropriateness" of CT scans ordered. This last point can be measured in a variety of ways, such as the percentage of low-risk patients (as defined by decision-support) receiving CT, as well as the diagnostic yield of the CTs that are ordered.

Procedure:

This study will be supported by several strategies including the integration of decision-support into CT ordering procedures in consultation with participating sites. This will also be supported by a voluntary pre-intervention Physician Survey to measure knowledge and attitudes towards CT ordering and decision-support, as well as the perceived barriers to implementing decision-support in their practice. Finally, throughout the intervention physicians and sites will be provided with "audit and feedback" (clinical informatics) on their CT ordering practices in relation to their peers. This feedback will be provided through existing AHS data systems through the Department of Data Integration, Measurement, and Reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patients: All patients presenting to pre-determined Alberta emergency departments with head injuries and suspected pulmonary embolism will be targeted for evaluation of CT appropriateness. For the CT Head, patients >16 with a CEDIS Triage code of "Head Injury" will be eligible. For the CT Pulmonary Angiography (CTPA) patients age 18-85 with CEDIS Triage codes of "Chest Pain (Noncardiac Features)", "Shortness of Breath", or "Syncope/Presyncope" will be eligible.
* Health Professionals: Engagement in this project will fall within the professional responsibilities and mandate for many if not all of these individuals will be supported by zone leadership in each domain. The interventions proposed are educational and voluntary in nature; as there are clinical situations in which clinical judgement is expected to supersede clinical guidelines, and therefore no coercive measures will be taken to impose universal physician compliance.

Exclusion Criteria:

* Patients under 16 years of age for CT head, under 18 or over 85 years of age for CT pulmonary angiography.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52058 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mild traumatic brain injury who undergo a CT head | All presenting patients for a period of 30 months (15 months pre-intervention administrative data, and 15 months of administrative date during the intervention)/
Proportion of patients with suspected Pulmonary Embolism who undergo a CTPA scan | All presenting patients for a period of 30 months (15 months pre-intervention administrative data, and 15 months of administrative date during the intervention)

SECONDARY OUTCOMES:
Proportion of patients with mild traumatic brain injury who undergo a CT Head for which a CT Head is recommended by the Canadian CT Head Rule | All presenting patients for a period of 30 months (15 months pre-intervention administrative data, and 15 months of administrative date during the intervention)
Proportion of patients with suspected pulmonary embolism who undergo a CTPA scan for which a CTPA scan is recommended after applying the Well's Score, the Pulmonary Embolism Rule-Out Criteria (PERC), and receiving D-Dimer test results. | All presenting patients for a period of 30 months (15 months pre-intervention administrative data, and 15 months of administrative date during the intervention)
Proportion of patients who return to the ED within 30 days with the same presenting complaint and undergo a CT Head or CTPA | Patients will be followed from presentation to the ED up until 30 days post-discharge from the ED

CONTACTS AND LOCATIONS:
Overall Officials: Eddy S. Lang, MD, Principal Investigator — University of Calgary; Andrew McRae, MD, Study Director — University of Calgary; James Andruchow, MD, Study Director — University of Calgary; Grant Innes, MD, Study Director — University of Calgary
Locations (16):
- Canada (16):
  - Foothills Medical Centre - C231, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Sheldom M. Chumir Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Grey Nuns CommunityHospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmontyon, Alberta
  - Northern Lights Regional Hospital, Fort McMurray, Alberta
  - Fort Saskatchewan Health Centre, Ft Saskatchewan, Alberta
  - Queen Elizabeth II Hospital, Grande Prairie, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - Strathcona Community Hospital, Sherwood Park, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta

REFERENCES:
- [Background] Kocher KE, Meurer WJ, Fazel R, Scott PA, Krumholz HM, Nallamothu BK. National trends in use of computed tomography in the emergency department. Ann Emerg Med. 2011 Nov;58(5):452-62.e3. doi: 10.1016/j.annemergmed.2011.05.020. Epub 2011 Aug 11. PMID 21835499
- [Background] Baker LC, Atlas SW, Afendulis CC. Expanded use of imaging technology and the challenge of measuring value. Health Aff (Millwood). 2008 Nov-Dec;27(6):1467-78. doi: 10.1377/hlthaff.27.6.1467. PMID 18997202
- [Background] Studdert DM, Mello MM, Sage WM, DesRoches CM, Peugh J, Zapert K, Brennan TA. Defensive medicine among high-risk specialist physicians in a volatile malpractice environment. JAMA. 2005 Jun 1;293(21):2609-17. doi: 10.1001/jama.293.21.2609. PMID 15928282
- [Background] Schattner A. Angst-driven medicine? QJM. 2009 Jan;102(1):75-8. doi: 10.1093/qjmed/hcn164. PMID 19095678
- [Background] Bishop TF, Federman AD, Keyhani S. Physicians' views on defensive medicine: a national survey. Arch Intern Med. 2010 Jun 28;170(12):1081-3. doi: 10.1001/archinternmed.2010.155. No abstract available. PMID 20585077
- [Background] Miller P, Kendrick D, Bentley E, Fielding K. Cost-effectiveness of lumbar spine radiography in primary care patients with low back pain. Spine (Phila Pa 1976). 2002 Oct 15;27(20):2291-7. doi: 10.1097/00007632-200210150-00021. PMID 12394910
- [Background] Berdahl CT, Vermeulen MJ, Larson DB, Schull MJ. Emergency department computed tomography utilization in the United States and Canada. Ann Emerg Med. 2013 Nov;62(5):486-494.e3. doi: 10.1016/j.annemergmed.2013.02.018. Epub 2013 May 14. PMID 23683773
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Brenner DJ, Hricak H. Radiation exposure from medical imaging: time to regulate? JAMA. 2010 Jul 14;304(2):208-9. doi: 10.1001/jama.2010.973. No abstract available. PMID 20628137
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] Stiell IG, Greenberg GH, McKnight RD, Nair RC, McDowell I, Reardon M, Stewart JP, Maloney J. Decision rules for the use of radiography in acute ankle injuries. Refinement and prospective validation. JAMA. 1993 Mar 3;269(9):1127-32. doi: 10.1001/jama.269.9.1127. PMID 8433468
- [Background] Stiell IG, Greenberg GH, Wells GA, McDowell I, Cwinn AA, Smith NA, Cacciotti TF, Sivilotti ML. Prospective validation of a decision rule for the use of radiography in acute knee injuries. JAMA. 1996 Feb 28;275(8):611-5. PMID 8594242
- [Background] Hoffman JR, Mower WR, Wolfson AB, Todd KH, Zucker MI. Validity of a set of clinical criteria to rule out injury to the cervical spine in patients with blunt trauma. National Emergency X-Radiography Utilization Study Group. N Engl J Med. 2000 Jul 13;343(2):94-9. doi: 10.1056/NEJM200007133430203. PMID 10891516
- [Background] Stiell IG, Wells GA, Vandemheen KL, Clement CM, Lesiuk H, De Maio VJ, Laupacis A, Schull M, McKnight RD, Verbeek R, Brison R, Cass D, Dreyer J, Eisenhauer MA, Greenberg GH, MacPhail I, Morrison L, Reardon M, Worthington J. The Canadian C-spine rule for radiography in alert and stable trauma patients. JAMA. 2001 Oct 17;286(15):1841-8. doi: 10.1001/jama.286.15.1841. PMID 11597285
- [Background] Kuppermann N, Holmes JF, Dayan PS, Hoyle JD Jr, Atabaki SM, Holubkov R, Nadel FM, Monroe D, Stanley RM, Borgialli DA, Badawy MK, Schunk JE, Quayle KS, Mahajan P, Lichenstein R, Lillis KA, Tunik MG, Jacobs ES, Callahan JM, Gorelick MH, Glass TF, Lee LK, Bachman MC, Cooper A, Powell EC, Gerardi MJ, Melville KA, Muizelaar JP, Wisner DH, Zuspan SJ, Dean JM, Wootton-Gorges SL; Pediatric Emergency Care Applied Research Network (PECARN). Identification of children at very low risk of clinically-important brain injuries after head trauma: a prospective cohort study. Lancet. 2009 Oct 3;374(9696):1160-70. doi: 10.1016/S0140-6736(09)61558-0. Epub 2009 Sep 14. PMID 19758692
- [Background] Osmond MH, Klassen TP, Wells GA, Correll R, Jarvis A, Joubert G, Bailey B, Chauvin-Kimoff L, Pusic M, McConnell D, Nijssen-Jordan C, Silver N, Taylor B, Stiell IG; Pediatric Emergency Research Canada (PERC) Head Injury Study Group. CATCH: a clinical decision rule for the use of computed tomography in children with minor head injury. CMAJ. 2010 Mar 9;182(4):341-8. doi: 10.1503/cmaj.091421. Epub 2010 Feb 8. PMID 20142371
- [Background] Stiell IG, Wells GA, Vandemheen K, Clement C, Lesiuk H, Laupacis A, McKnight RD, Verbeek R, Brison R, Cass D, Eisenhauer ME, Greenberg G, Worthington J. The Canadian CT Head Rule for patients with minor head injury. Lancet. 2001 May 5;357(9266):1391-6. doi: 10.1016/s0140-6736(00)04561-x. PMID 11356436
- [Background] Stiell IG, Clement CM, Rowe BH, Schull MJ, Brison R, Cass D, Eisenhauer MA, McKnight RD, Bandiera G, Holroyd B, Lee JS, Dreyer J, Worthington JR, Reardon M, Greenberg G, Lesiuk H, MacPhail I, Wells GA. Comparison of the Canadian CT Head Rule and the New Orleans Criteria in patients with minor head injury. JAMA. 2005 Sep 28;294(12):1511-8. doi: 10.1001/jama.294.12.1511. PMID 16189364
- [Background] Harnan SE, Pickering A, Pandor A, Goodacre SW. Clinical decision rules for adults with minor head injury: a systematic review. J Trauma. 2011 Jul;71(1):245-51. doi: 10.1097/TA.0b013e31820d090f. PMID 21818031
- [Background] Wells PS, Anderson DR, Rodger M, Stiell I, Dreyer JF, Barnes D, Forgie M, Kovacs G, Ward J, Kovacs MJ. Excluding pulmonary embolism at the bedside without diagnostic imaging: management of patients with suspected pulmonary embolism presenting to the emergency department by using a simple clinical model and d-dimer. Ann Intern Med. 2001 Jul 17;135(2):98-107. doi: 10.7326/0003-4819-135-2-200107170-00010. PMID 11453709
- [Background] Kline JA, Courtney DM, Kabrhel C, Moore CL, Smithline HA, Plewa MC, Richman PB, O'Neil BJ, Nordenholz K. Prospective multicenter evaluation of the pulmonary embolism rule-out criteria. J Thromb Haemost. 2008 May;6(5):772-80. doi: 10.1111/j.1538-7836.2008.02944.x. Epub 2008 Mar 3. PMID 18318689
- [Background] Ceriani E, Combescure C, Le Gal G, Nendaz M, Perneger T, Bounameaux H, Perrier A, Righini M. Clinical prediction rules for pulmonary embolism: a systematic review and meta-analysis. J Thromb Haemost. 2010 May;8(5):957-70. doi: 10.1111/j.1538-7836.2010.03801.x. Epub 2010 Feb 2. PMID 20149072
- [Background] Goldhaber SZ, Bounameaux H. Pulmonary embolism and deep vein thrombosis. Lancet. 2012 May 12;379(9828):1835-46. doi: 10.1016/S0140-6736(11)61904-1. Epub 2012 Apr 10. PMID 22494827
- [Background] Singh B, Parsaik AK, Agarwal D, Surana A, Mascarenhas SS, Chandra S. Diagnostic accuracy of pulmonary embolism rule-out criteria: a systematic review and meta-analysis. Ann Emerg Med. 2012 Jun;59(6):517-20.e1-4. doi: 10.1016/j.annemergmed.2011.10.022. Epub 2011 Dec 15. PMID 22177109
- [Background] Hayward RS, Guyatt GH, Moore KA, McKibbon KA, Carter AO. Canadian physicians' attitudes about and preferences regarding clinical practice guidelines. CMAJ. 1997 Jun 15;156(12):1715-23. PMID 9220923
- [Background] Graham ID, Stiell IG, Laupacis A, O'Connor AM, Wells GA. Emergency physicians' attitudes toward and use of clinical decision rules for radiography. Acad Emerg Med. 1998 Feb;5(2):134-40. doi: 10.1111/j.1553-2712.1998.tb02598.x. PMID 9492134
- [Background] Eagles D, Stiell IG, Clement CM, Brehaut J, Taljaard M, Kelly AM, Mason S, Kellermann A, Perry JJ. International survey of emergency physicians' awareness and use of the Canadian Cervical-Spine Rule and the Canadian Computed Tomography Head Rule. Acad Emerg Med. 2008 Dec;15(12):1256-61. doi: 10.1111/j.1553-2712.2008.00265.x. Epub 2008 Oct 17. PMID 18945241
- [Background] Melnick ER, Szlezak CM, Bentley SK, Dziura JD, Kotlyar S, Post LA. CT overuse for mild traumatic brain injury. Jt Comm J Qual Patient Saf. 2012 Nov;38(11):483-9. doi: 10.1016/s1553-7250(12)38064-1. PMID 23173394
- [Background] Stiell IG, Clement CM, Grimshaw JM, Brison RJ, Rowe BH, Lee JS, Shah A, Brehaut J, Holroyd BR, Schull MJ, McKnight RD, Eisenhauer MA, Dreyer J, Letovsky E, Rutledge T, Macphail I, Ross S, Perry JJ, Ip U, Lesiuk H, Bennett C, Wells GA. A prospective cluster-randomized trial to implement the Canadian CT Head Rule in emergency departments. CMAJ. 2010 Oct 5;182(14):1527-32. doi: 10.1503/cmaj.091974. Epub 2010 Aug 23. PMID 20732978
- [Background] Graham ID, Stiell IG, Laupacis A, McAuley L, Howell M, Clancy M, Durieux P, Simon N, Emparanza JI, Aginaga JR, O'connor A, Wells G. Awareness and use of the Ottawa ankle and knee rules in 5 countries: can publication alone be enough to change practice? Ann Emerg Med. 2001 Mar;37(3):259-66. doi: 10.1067/mem.2001.113506. PMID 11223761
- [Background] Brehaut JC, Stiell IG, Visentin L, Graham ID. Clinical decision rules "in the real world": how a widely disseminated rule is used in everyday practice. Acad Emerg Med. 2005 Oct;12(10):948-56. doi: 10.1197/j.aem.2005.04.024. Epub 2005 Sep 15. PMID 16166599
- [Background] Brehaut JC, Stiell IG, Graham ID. Will a new clinical decision rule be widely used? The case of the Canadian C-spine rule. Acad Emerg Med. 2006 Apr;13(4):413-20. doi: 10.1197/j.aem.2005.11.080. Epub 2006 Mar 10. PMID 16531607
- [Background] van Ravesteijn H, van Dijk I, Darmon D, van de Laar F, Lucassen P, Olde Hartman T, van Weel C, Speckens A. The reassuring value of diagnostic tests: a systematic review. Patient Educ Couns. 2012 Jan;86(1):3-8. doi: 10.1016/j.pec.2011.02.003. Epub 2011 Mar 6. PMID 21382687
- [Background] Curran JA, Brehaut J, Patey AM, Osmond M, Stiell I, Grimshaw JM. Understanding the Canadian adult CT head rule trial: use of the theoretical domains framework for process evaluation. Implement Sci. 2013 Feb 21;8:25. doi: 10.1186/1748-5908-8-25. PMID 23433082
- [Background] Ranmuthugala G, Plumb JJ, Cunningham FC, Georgiou A, Westbrook JI, Braithwaite J. How and why are communities of practice established in the healthcare sector? A systematic review of the literature. BMC Health Serv Res. 2011 Oct 14;11:273. doi: 10.1186/1472-6963-11-273. PMID 21999305
- [Background] Fung-Kee-Fung M, Watters J, Crossley C, Goubanova E, Abdulla A, Stern H, Oliver TK. Regional collaborations as a tool for quality improvements in surgery: a systematic review of the literature. Ann Surg. 2009 Apr;249(4):565-72. doi: 10.1097/SLA.0b013e31819ec608. PMID 19300234
- [Background] Li LC, Grimshaw JM, Nielsen C, Judd M, Coyte PC, Graham ID. Use of communities of practice in business and health care sectors: a systematic review. Implement Sci. 2009 May 17;4:27. doi: 10.1186/1748-5908-4-27. PMID 19445723
- [Background] Barnett S, Jones SC, Bennett S, Iverson D, Bonney A. General practice training and virtual communities of practice - a review of the literature. BMC Fam Pract. 2012 Aug 21;13:87. doi: 10.1186/1471-2296-13-87. PMID 22905827
- [Background] Perry JJ, Stiell IG. Impact of clinical decision rules on clinical care of traumatic injuries to the foot and ankle, knee, cervical spine, and head. Injury. 2006 Dec;37(12):1157-65. doi: 10.1016/j.injury.2006.07.028. Epub 2006 Oct 31. PMID 17078955
- [Background] Stiell IG, Clement CM, Grimshaw J, Brison RJ, Rowe BH, Schull MJ, Lee JS, Brehaut J, McKnight RD, Eisenhauer MA, Dreyer J, Letovsky E, Rutledge T, MacPhail I, Ross S, Shah A, Perry JJ, Holroyd BR, Ip U, Lesiuk H, Wells GA. Implementation of the Canadian C-Spine Rule: prospective 12 centre cluster randomised trial. BMJ. 2009 Oct 29;339:b4146. doi: 10.1136/bmj.b4146. PMID 19875425
- [Background] Atkins D, Best D, Briss PA, Eccles M, Falck-Ytter Y, Flottorp S, Guyatt GH, Harbour RT, Haugh MC, Henry D, Hill S, Jaeschke R, Leng G, Liberati A, Magrini N, Mason J, Middleton P, Mrukowicz J, O'Connell D, Oxman AD, Phillips B, Schunemann HJ, Edejer T, Varonen H, Vist GE, Williams JW Jr, Zaza S; GRADE Working Group. Grading quality of evidence and strength of recommendations. BMJ. 2004 Jun 19;328(7454):1490. doi: 10.1136/bmj.328.7454.1490. PMID 15205295
- [Background] Grafstein E, Bullard MJ, Warren D, Unger B; CTAS National Working Group. Revision of the Canadian Emergency Department Information System (CEDIS) Presenting Complaint List version 1.1. CJEM. 2008 Mar;10(2):151-73. doi: 10.1017/s1481803500009878. No abstract available. English, French. PMID 18371253
- [Background] Campbell MK, Thomson S, Ramsay CR, MacLennan GS, Grimshaw JM. Sample size calculator for cluster randomized trials. Comput Biol Med. 2004 Mar;34(2):113-25. doi: 10.1016/S0010-4825(03)00039-8. PMID 14972631
- [Background] Boyle A, Santarius L, Maimaris C. Evaluation of the impact of the Canadian CT head rule on British practice. Emerg Med J. 2004 Jul;21(4):426-8. PMID 15208223
- [Background] Sodickson A, Baeyens PF, Andriole KP, Prevedello LM, Nawfel RD, Hanson R, Khorasani R. Recurrent CT, cumulative radiation exposure, and associated radiation-induced cancer risks from CT of adults. Radiology. 2009 Apr;251(1):175-84. doi: 10.1148/radiol.2511081296. PMID 19332852
- [Derived] Andruchow JE, Grigat D, McRae AD, Innes G, Vatanpour S, Wang D, Taljaard M, Lang E. Decision support for computed tomography in the emergency department: a multicenter cluster-randomized controlled trial. CJEM. 2021 Sep;23(5):631-640. doi: 10.1007/s43678-021-00170-3. Epub 2021 Aug 5. PMID 34351598